CLINICAL TRIAL: NCT01013428
Title: FLEX-Trial: Prospective Sonographic Assessment Of Healing Process Following Suture of Profound Flexor Tendon Due to Traumatic Rupture of FDP-Tendon in Zone II.
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Gustav Andreisek, md, University of Zurich
Other Study IDs: 001
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Tendon Injury
Keywords: Traumatic Rupture of Tendon
MeSH Terms: conditions — Tendon Injuries | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Ultrasound — Ultrasound will be used to evaluate tendons.

SUMMARY:
To prospectively assess the healing process following suture of profound fexor tendon due to traumatic rupture of FDP-Tendon in Zone II by ultrasound.

ELIGIBILITY:
Inclusion criteria:

* All patients with traumatic rupture of FDP-tendon in zone II.

Exclusion criteria:

* < 18years;
* Fracture;
* crush injury; (partial) amputation;
* RA;
* CPPD;
* CP;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland